CLINICAL TRIAL: NCT07271147
Title: The Effect of Dexmedetomidine Combined With Percutaneous Auricular Vagus Nerve Stimulation on Postoperative Nausea and Vomiting in Female Laparoscopic Patients: A Randomized Controlled Trial
Brief Title: Effects of taVNS Combined With Dexmedetomidine on POVN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Chaochao Zhong, Principal Investigator, Affiliated Hospital of Nantong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-K265-02
Record Dates: First submitted 2025-11-19; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine combined with taVNS(taVNS group) (Experimental): Patients in the taVNS group will have a transcutaneous auricular vagus nerve stimulation device with a transparent, non-insulated thin film placed on the cymba conchae of the left ear. TaVNS will be administered on the day of surgery (starting 30 minutes before anesthesia induction and continuing until the end of the surgery, terminating after the removal of the endotracheal tube in the PACU). The stimulation parameters are set as follows: frequency 25 Hz, pulse width 200 μs, 30 seconds on / 30 seconds off, with the current intensity set to the maximum amplitude the patient can tolerate (just below the pain threshold).
  Dexmedetomidine was administered intravenously by infusion pump (0.5 μg/kg over 10 minutes, followed by continuous infusion at 0.4 μg/kg/h) in combination with taVNS (initiated 30 minutes before anesthesia induction and terminated after tracheal tube removal in the PACU upon the conclusion of the surgery).
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulator; Drug: Dexmedetomidine
- Dexmedetomidine combined with sham transcutaneous auricular vagus nerve stimulation (Sham Comparator): Patients in the Sham taVNS group will have a transcutaneous auricular vagus nerve stimulation device with a transparent insulating film placed on the cymba conchae of the left ear on the day of surgery. The stimulation parameters, method, and duration will be the same as those in the taVNS group. However, due to the insulating film applied to the stimulation device in the sham group, patients will not actually receive any stimulation.
  Dexmedetomidine was administered intravenously by infusion pump (0.5 μg/kg over 10 minutes, followed by continuous infusion at 0.4 μg/kg/h) in combination with taVNS (initiated 30 minutes before anesthesia induction and terminated after tracheal tube removal in the PACU upon the conclusion of the surgery).
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulator — Intervention Timing of Transcutaneous Auricular Vagus Nerve Stimulator: The intervention will begin 30 minutes before anesthesia induction and continue until the end of the surgery, terminating after the removal of the endotracheal tube in the PACU. The stimulation parameters are set as follows: frequency 25 Hz, pulse width 200 μs, 30 seconds on / 30 seconds off, with the current intensity set to the maximum amplitude the patient can tolerate (just below the pain threshold).
  Arms: Dexmedetomidine combined with taVNS(taVNS group)
Drug: Dexmedetomidine — Dexmedetomidine was administered intravenously by infusion pump (0.5 μg/kg over 10 minutes, followed by continuous infusion at 0.4 μg/kg/h) in combination with taVNS (initiated 30 minutes before anesthesia induction and terminated after tracheal tube removal in the PACU upon the conclusion of the surgery).

SUMMARY:
To explore the effects and possible mechanisms of dexmedetomidine combined with taVNS on the incidence of postoperative nausea and vomiting in female patients undergoing laparoscopic surgery

DETAILED DESCRIPTION:
Patients are recruited one week prior to the start of the trial, during which they are informed about the experimental protocol and associated risks. After obtaining informed consent and signatures, they are enrolled as study participants. Patients who meet the trial criteria are randomly assigned in a 1:1 ratio to the control group (sham taVNS group) and the intervention group (taVNS group, with taVNS intervention starting 30 minutes prior to anesthesia induction and continuing until the end of surgery, terminating after the removal of the endotracheal tube in the PACU), in a double-blind manner (with taVNS intervention and postoperative follow-up conducted by different researchers).

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 to 65;
* Elective laparoscopic surgery under general anesthesia;
* Classified as American Society of Anesthesiologists (ASA) physical status I to II;
* Capable of understanding the study procedures and various assessment scales and able to effectively communicate with the researchers;
* Willing to participate in the study and provide written informed consent.

Exclusion Criteria:

* Patients with ASA anesthesia classification ≥ III;
* Poorly controlled hypertension, atrioventricular block ≥ second degree, obesity (BMI > 30 kg/m²);
* Pregnant or breastfeeding;
* Known allergy to drugs used in the study protocol, history of traumatic brain injury, history of gastrointestinal surgery;
* Liver or kidney dysfunction (liver enzymes or creatinine ≥ 1.5 times the normal value), alcoholism or drug abuse, mental illness, use of antiemetics, opioids, psychoactive drugs, or corticosteroids within 24 hours before surgery;
* Patients with implanted stimulators (such as pacemakers, implantable vagus nerve stimulators, deep brain stimulators, spinal cord stimulators, etc.), cochlear implants, or metal implants (except in dental cases);
* Skin lesions or dermatological diseases at the site of electrical stimulation;
* Preoperative heart rate < 50 bpm or the presence of sinoatrial node disease or second-degree or higher atrioventricular block;
* Patients unable to cooperate with assessments;
* Patients participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2025-11-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative PONV | The first 24 hours postoperatively
  Patients who experience at least one episode of nausea, vomiting, or retching, or any combination of these, within the first 24 hours after surgery are considered to have PONV.

SECONDARY OUTCOMES:
The frequency of nausea, retching and vomiting within 2 hours, 6 hours, 24 hours and 48 hours after surgery. | From 2 hours postoperatively to 48 hours postoperatively
  Postoperative nausea is defined as the occurrence of nausea at least once without retching or vomiting. Retching is defined as the patient experiencing regular spasms in the chest and abdominal muscles without the expulsion of gastric contents. Vomiting is defined as vomiting or retching at least once.
Frequency of remedial antiemetic administration within 2 hours, 6 hours, 24 hours and 48 hours after surgery. | From 2 hours postoperatively to 48 hours postoperatively
The severity of nausea and vomiting within 2 hours, 6 hours, 24 hours and 48 hours after surgery. | From 2 hours postoperatively to 48 hours postoperatively
  Severity was assessed using a 4-point Likert scale: 0 = none, 1 = mild, 2 = moderate, 3 = severe.
Incidence of PONV at 2 hours, 6 hours, and 48 hours postoperatively | From 2 hours postoperatively to 48 hours postoperatively
  Patients who experienced at least one episode of nausea, vomiting, retching, or any combination thereof within the first 2, 6, or 48 hours after surgery were considered to have PONV.
Postoperative NRS pain scores at 2 h, 6 h, 24 h, and 48 h | From 2 hours postoperatively to 48 hours postoperatively
  The NRS (Numerical Rating Scale) is used to assess the intensity of pain.Minimum: 0 Maximum: 10.The higher the score, the more severe the pain.
Number of patient-controlled analgesia (PCA) pump activations at 2 h, 6 h, 24 h, and 48 h after surgery | From 2 hours postoperatively to 48 hours postoperatively
Frequency of rescue analgesic use at 2 h, 6 h, 24 h, and 48 h postoperatively | From 2 hours postoperatively to 48 hours postoperatively
Intraoperative incidence of hypotension and bradycardia | during surgery
  Hypotension was defined as a mean arterial pressure < 60 mmHg, and bradycardia as a heart rate < 50 bpm.
Incidence of other adverse reactions within 48 h after surgery (dizziness, somnolence, dry mouth, skin irritation). | The first 48 hours postoperatively
Preoperative and 24-hour postoperative Hospital Anxiety and Depression Scale (HADS) | From 1 day preoperatively to 24 hours postoperatively
  The Hospital Anxiety and Depression Scale (HADS) is used to assess the severity of anxiety and depression in individuals.
  Full scale title: Hospital Anxiety and Depression Scale (HADS) - Full 14-Item Version Minimum score: 0 Maximum score: 42 (0-21 for the anxiety subscale and 0-21 for the depression subscale) Interpretation: Higher scores indicate greater severity of anxiety and/or depression, representing worse outcomes.
PROMIS SD-SF 8a Assessment on Preoperative and 24-hour Postoperative | From 1 day preoperatively to 24 hours postoperatively
  The Patient-Reported Outcomes Measurement Information System Sleep Disturbance - Short Form 8a (PROMIS SD-SF 8a) is an 8-item self-reported questionnaire developed by the Patient-Reported Outcomes Measurement Information System to assess sleep disturbance over the past 7 days. It evaluates aspects such as difficulty falling asleep, sleep maintenance, sleep quality, and daytime functioning, providing a standardized measure of sleep disturbance severity.
  Full scale title Patient-Reported Outcomes Measurement Information System Sleep Disturbance Short Form 8a (PROMIS SD-SF 8a) - 8-Item Version Score range Minimum: 8 Maximum: 40 Interpretation Higher scores indicate greater sleep disturbance over the past seven days, corresponding to worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Chao Zhong, Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No